CLINICAL TRIAL: NCT02310555
Title: Prospective Randomised Study Comparing Surgical Techniques in Patients With Diabetes Mellitus-II And Obesity
Brief Title: Surgical Techniques in Diabetes Mellitus-II and Obesity. Metabolic Surgery Study (MSS)
Acronym: MSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Juan Lujan, Section chief, Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCUVA-MSS-JL
Record Dates: First submitted 2014-11-26; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus; Obesity
Keywords: Metabolic surgery
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gastric bypass (Active Comparator): classic Gastric bypass
  Interventions: Procedure: Gastric bypass
- Modified gastric bypass. (Active Comparator): Modified gastric bypass. Resection body and fundus gastric
  Interventions: Procedure: Modified gastric bypass.
- Slevee Gastrectomy (Active Comparator): Slevee Gastrectomy
  Interventions: Procedure: Slevee Gastrectomy

INTERVENTIONS:
Procedure: Gastric bypass
  Arms: Gastric bypass
Procedure: Modified gastric bypass.
  Arms: Modified gastric bypass.
Procedure: Slevee Gastrectomy
  Arms: Slevee Gastrectomy

SUMMARY:
The aim of this study is to compare clinical and laboratory findings of three surgical techniques in metabolic surgery in patients with type II diabetes mellitus and obesity (BMI> 30).

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-40
* Diabetes Mellitus type II less than 10 years of evolution.
* Anti-GAD, anti-pancreatic islets negative antibodies.
* C peptide normally between 0.9 and 4.
* Glycosylated hemoglobin greater than 6.5%.
* Less than 5 years of use insulin.

Exclusion Criteria:

* Cirrosis hepática.
* coagulopathies.
* Type 1 diabetes.
* HIV positive.
* Stomach or small intestine previous surgeries .
* Diseases of the exocrine pancreas: pancreatitis, pancreatectomy, neoplasia, cystic fibrosis, hemochromatosis.
* Endocrinopathies: acromegaly, glucagonoma, Cushing's syndrome, pheochromocytoma, hyperthyroidism, somatostatinoma, aldosteronoma.
* Genetic syndromes with diabetes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Remission diabetes mellitus type II | Durign two years
  1. Partial remission: Not diagnostic of DM HbA1c (<6.5%); Basal glucose 100-125 mg / dl (5.6-6.9 mmol / l); Absence of drug treatment; At least one year.
  2. Complete remission: Normal HbA1c (<6%); basal glucose <100 mg / dl (<5.6 mmol / l); Absence of drug treatment; At least one year.
  3. Prolonged remission: At least 5 years of remission.
  4. Improvement: HbA1c <7% with pharmacological treatment.

SECONDARY OUTCOMES:
Weight loss | During two years
Adverse effects in the short term | During three months since surgery
  We'll measure the number of patients with postoperative complications and the the degree of severity of Clavien- Dindo Classification
Adverse effects in the long term | Since third month after surgery untiil two years
  We'll measure the number of patients with postoperative complications and the the degree of severity of Clavien- Dindo Classification

CONTACTS AND LOCATIONS:
Overall Officials: Juan A. Luján Mompean, Ph D; Section chief, Principal Investigator — Hospital Clínico Universitario Virgen Arrixaca
Locations (1):
- Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia, Spain